CLINICAL TRIAL: NCT01176318
Title: A Double Blind, Placebo Controlled Multicentre Study of the Effects of Standard Care Plus Erdosteine (Erdotin) Versus Standard Care Plus Placebo on Cough in Acute Exacerbations of Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Erdosteine (Erdotin) Versus Standard Care Plus Placebo on Erdosteine for Treatment of Cough in Acute Exacerbations of Chronic Obstructive Pulmonary Disease (COPD)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: grant was withdrawn no financial support to conduct the study.
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: Galen Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Erd090908
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: cough; exacerbation; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cough | interventions — erdosteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- erdosteine (Experimental): standard care plus erdosteine for 10 days
  Interventions: Drug: Erdosteine
- placebo (Placebo Comparator): Standard care for exacerbation of COPD plus placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erdosteine — capsule 300mg twice daily for 10 days
  Other Names: erdotin
  Arms: erdosteine
Drug: Placebo — placebo capsule, twice daily for 10 days
  Arms: placebo

SUMMARY:
This is a parallel group, double-blind, placebo controlled, multi-centre, randomised trial.

60 patients to be included who are adult patients admitted to hospital with a clinical diagnosis of acute exacerbation of Chronic Obstructive Pulmonary Disease (COPD). Acute exacerbation of COPD will be defined as sustained worsening of the patient's condition with an increase in cough and one or more of dyspnoea, sputum volume or sputum purulence, necessitating a change in regular medication.

The primary objective of this study is to evaluate the effectiveness of standard care plus erdosteine in reducing hourly cough (24 hour cough recording using automated cough recorder) measured from baseline (Day 0) and at Day 5 of treatment, compared with standard care plus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male/females aged between 40-80 years
* Previous diagnosis of COPD
* Acute exacerbation of COPD requiring treatment with antibiotics and/or corticosteroids
* Symptoms of increased breathlessness, cough, sputum volume or sputum purulence
* Acute exacerbation of COPD hospitalised within 24hrs of study participation.
* On a stable therapeutic regimen for COPD for 8 weeks prior to inclusion
* Known history of cigarette smoking at least 10 pack yrs
* Willing and able to comply with study procedures
* Able to provide written informed consent to participate

Exclusion Criteria:

* Acute exacerbation of COPD within 8 weeks prior to inclusion
* Arterial blood gas on admission < pH 7.26
* Currently on treatment with mucolytics
* Patients suffering from post nasal drip, or gastro-oesophageal reflux disease
* Clinically significant or unstable concurrent disease e.g. left ventricular failure, diabetes mellitus
* On long-term oxygen therapy
* Known or suspected hypersensitivity to erdosteine

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08-10 (Estimated); Primary Completion 2011-10-12 (Estimated); Study Completion 2012-01-13 (Estimated)

PRIMARY OUTCOMES:
24 hr cough recording | 5 days
  The primary objective is to evaluate the effectiveness of standard care plus erdosteine in reducing hourly cough (24 hour cough recording using automated cough recorder) measureing differerrence in hourly cough rate from baseline (Day 0) and Day 5 of treatment, compared with standard care plus placebo

SECONDARY OUTCOMES:
Quality of life questionnaire | 10 days
  QOL questionnaire score,Compare differece in scores recorded at baseline (day 0) and day 10, compare the difference between erdosteine plus standard care with that of standard care plus placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Alyn H Morice, FRCP, Principal Investigator — Hull and east Yorkshire NHS trust
Locations (1):
- Castle Hill Hospital, Cottingham, East Yorkshire, United Kingdom